CLINICAL TRIAL: NCT04155905
Title: Fistulotomy Versus Fistulotomy With Marsupialization of Wound Edges in Simple Perianal Fistula, a Comparative Clinical Trial
Brief Title: Marsupialization of Anal Fistulotomy Wound Accelerates Healing and Decreases Post Operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: marsupialization anal fistula
Record Dates: First submitted 2019-11-02; First posted 2019-11-07 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Anal Fistula
Keywords: simple anal fistula; marsupialization
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: comparison between two groups of patients with simple anal fistula subjected to different types of treatment
Who Masked: Participant
Masking Description: patients don't know the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A fistulotomy group (Active Comparator): 35 patients with simple anal fistula subjected to fistulotomy
  Interventions: Procedure: fistulotomy
- group B marsupialization group (Active Comparator): 35 patients with simple anal fistula subjected to fistulotomy and marsupialization of fistulotomy wound
  Interventions: Procedure: fistulotomy and marsupialization of wound edges

INTERVENTIONS:
Procedure: fistulotomy and marsupialization of wound edges — after defining the fistulous track it was laid open (marsupialization) was done together with marsupialization of the wound edge with vicryl 3\0 sutures
  Arms: group B marsupialization group
Procedure: fistulotomy — after defining the fistulous track it was laid open (marsupialization)
  Arms: group A fistulotomy group

SUMMARY:
comparison between to groups of patients with simple anal fistula one group underwent sistulotomy the other underwent fistulotomy and marsupialization of the wound edges , the investigator tested the incidence of postoperative complications , time of wound healing , operative time

DETAILED DESCRIPTION:
This randomized controlled trial was carried in the period between May 2018 and April 2019, on 70 patients undergoing fistulotomy for treatment of simple perianal fistula. Patients were randomly allocated into two equal groups each 35 patients, group A; underwent fistulotomy without marsupialization of the edges of fistulotomy wound. And group B; underwent fistulotomy with marsupialization of the wound edges.

Patients included in this study are those suffering simple non recurrent perianal fistula with ASA I and II.

the investigator excluded patients with secondary anal fistula, complex fistula, anal incontinence, previous anal surgery and any disease or drug that affects wound healing.

All patients were subjected to thorough history taking and careful anal examination to assess the sphincter integrity, define the fistulous track and internal opening, endo anal ultrasound or magnetic resonance imaging was ordered when needed.

Fistulotomy was done under spinal anesthesia in the lithotomy position after skin preparation and patient draping; anal examination under anesthesia was done, identification of the internal opening carried out using palpation and inspection using proctoscope, injection of hydrogen peroxide in the external opening done if internal opening couldn't be defined easily, then the fistulous track was probed, it was laid open using diathermy, in group B the wounds was marsupialized by suturing the skin edges to the edges of the track floor using absorbable sutures (polygalactin) 3\0. Figures (1) and (2) shows the probed fistulous track and its' wound after marsupialization.

Postoperative non adherent dressing impregnated with local anesthetic cream was applied to the wound.

Nonsteroidal analgesic injection was given in injection form as per need. Follow up was carried out in outpatient clinic by the study surgeons, patients who agreed for participation in the study was instructed to visit the clinic every week for the first three post-operative months then every month for the next 3 months and lastly two visits after 3 and 6 months, the attending surgeon records follow up data including status of wound healing, anal continence and fistula recurrence.

An informed written consent was taken from all study participants. Randomization was done using computer program. The study was approved from institutional review board and the ethical committee from our university.

Demographic data, operative data, and postoperative data including pain, post-operative complications and time taken for complete wound healing were collected, properly analyzed using the paired t test and Z test using SPSS program.

ELIGIBILITY:
Inclusion Criteria:

* Simple non recurrent perianal fistula with ASA I and II.

Exclusion Criteria:

* secondary anal fistula,
* complex fistula,
* anal incontinence,
* previous anal surgery
* Any disease or drug that affects wound healing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
operative time in minutes | intraoperative
  the time taken for completion of the procedure from fistulous track identification to the end of fistulotomy or marsupialization
postoperative pain using visual analogue scale | 1 week
  pain in the postoperative period
postoperative complications measured by clinical examination and anal sphincter manometry | 1 year
  examination of the patient for fistula recurrence, history, clinical examination and anal sphincter manometry for anal incontinence
wound healing time | 1 year
  time taken for wound to be completely healed

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided